CLINICAL TRIAL: NCT04208035
Title: Hepatitis C Elimination in the Netherlands (CELINE) - A National Multicenter Cohort Study Retrieving Lost to Follow-up Chronic Hepatitis C Patients
Brief Title: Hepatitis C Elimination in the Netherlands
Acronym: CELINE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Joost Drenth, Professor, MD, PhD, Radboud University Medical Center
Other Study IDs: 2018-4503
Record Dates: First submitted 2019-12-06; First posted 2019-12-23 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Chronic Hepatitis c
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of CELINE is to retrieve and re-evaluate lost to follow-up chronic hepatitis C patients in the Netherlands.

ELIGIBILITY:
Inclusion Criteria:

* Ever diagnosed with (possible) chronic HCV in the 15-year period prior to initiation of the study, defined as having had a positive anti-HCV or HCV RNA test
* Lost to follow-up, defined as the lack of a scheduled outpatient care appointment after the last known positive HCV test result

Exclusion Criteria:

* Younger than 18
* Deceased
* Not residing in the Netherlands
* Unknown current address
* Severe comorbidity or short life expectancy that limits patients from benefiting from retrieval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lost to follow-up (possibly) chronically HCV-infected patients
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2018-09-17 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of lost to follow-up (LTFU) patients successfully re-linked to care | End of study, on average 2.5 years after initiation

SECONDARY OUTCOMES:
Total number of LTFU patients in the investigated time period | 15 years prior to study initiation
Case ascertainment rate | End of study, on average 2.5 years after initiation
  Established contact (via telephone or in writing) with a patient who is eligible for retrieval
Awareness of HCV diagnosis among LTFU patients | End of study, on average 2.5 years after initiation
  Number of patients who were aware of their HCV diagnosis when they are invited for re-evaluation
Number of patients who never had an outpatient appointment with a hepatologist or infectious disease specialist after initial positive HCV test | End of study, on average 2.5 years after initiation
Number of viraemic patients at time of re-evaluation | End of study, on average 2.5 years after initiation
Liver fibrosis stage of retrieved patients | End of study, on average 2.5 years after initiation
Reasons for becoming LTFU | End of study, on average 2.5 years after initiation
Time of being LTFU | End of study, on average 2.5 years after initiation
  Defined as years since last (HCV-)related hospital visit
Mode of HCV transmission | End of study, on average 2.5 years after initiation
Sustained virological response | End of study, on average 2.5 years after initiation
  Defined as the absence of HCV RNA at least 12 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Joost Drenth, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Isfordink CJ, Brakenhoff SM, van Dijk M, van der Valk M, de Knegt RJ, Arends JE, Drenth JP; HepNed study group. Hepatitis C elimination in the Netherlands (CELINE): study protocol for nationwide retrieval of lost to follow-up patients with chronic hepatitis C. BMJ Open Gastroenterol. 2020 Apr 12;7(1):e000396. doi: 10.1136/bmjgast-2020-000396. eCollection 2020. PMID 32377367